CLINICAL TRIAL: NCT04024514
Title: Development of Renal Protection Protocol Using Low Dose Contrast Media and Spectral Computed Tomography in Chronic Kidney Disease Patients
Brief Title: Renal Protocol Protection in CKD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SNUH-2019-0343
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: HCC; CKD
Keywords: CT; Spectral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Experimental): Low CT contrast media dose
  Interventions: Other: low dose CT contrast media
- Standard dose (Active Comparator): Standard CT contrast media dose
  Interventions: Other: Standard dose CT contrast media

INTERVENTIONS:
Other: low dose CT contrast media — CT contrast media (Ioversol 320mgI/kg) is administrated at a dose of 300mgI/kg in low dose group
  Arms: Low dose
Other: Standard dose CT contrast media — CT contrast media (Ioversol 350mgI/kg) is administrated at a dose of 525mgI/kg in standard dose group.
  Arms: Standard dose

SUMMARY:
This study aims to investigate whether acceptable image quality is achievable using low contrast media dose and low keV imaging in chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* High risk group for developing HCC
* Scheduled contrast-enhanced CT for HCC diagnosis or surveillance
* chronic kidney disease (Estimated GFR < 60mL/min/1.73m2)

Exclusion Criteria:

* not a high risk group for developing HCC
* congestive hepatopathy
* on dialysis
* no venous access on forearm
* anticipated beam hardening artifact due to prosthesis
* relative/absolute contra-indication of contrast-enhanced CT except CKD (Estimated GFR < 60mL/min/1.73m2)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall image quality | 6 months after complete enrollment
  qualitative scoring for image quality on five-point scale (1: worst, 5: excellent, representative value is average score)

SECONDARY OUTCOMES:
Contrast media (CM) dose | 3 months after complete enrollment
  administered CM dose in each group
Incidence of Contrast media-induced nephrotoxicity | 3 days after contrast media administration
  serum Cr level increase by 25% or more of the baseline, or 0.5mg/dl in 3 days after contrast media administration without other cause
Image contrast | 12 months after complete enrollment
  qualitative scoring for image contrast on five-point scale (1: worst, 5: excellent, representative value is average score)
Lesion conspicuity | 12 months after complete enrollment
  qualitative scoring for focal lesion depiction on five-point scale
lesion (HCC) detection | 12 months after complete enrollment
  detection rate of focal liver lesion/HCC on CT

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon JH, Park JY, Lee SM, Lee ES, Kim JH, Lee JM. Renal protection CT protocol using low-dose and low-concentration iodine contrast medium in at-risk patients of HCC and with chronic kidney disease: a randomized controlled non-inferiority trial. Cancer Imaging. 2023 Oct 19;23(1):100. doi: 10.1186/s40644-023-00616-0. PMID 37858212